CLINICAL TRIAL: NCT06751368
Title: Aortic Valve Regurgitation After Surgical Repair for Subaortic Stenosis in Children
Brief Title: The Fate of Aortic Valve After SAS Surgery in Children
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2022-1727
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Subaortic Stenosis; Congenital Heart Disease; Aortic Regurgitation
MeSH Terms: conditions — Aortic Stenosis, Subvalvular; Heart Defects, Congenital; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Aortic valve regurgitation (AR) is a common complication following surgery for subaortic stenosis (SAS), yet the long-term outcomes and risk factors for postoperative significant AR (SAR) remain poorly understood. This study aims to investigate the incidence and risk factors of SAR in SAS patients and evaluate the long-term postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age from 0-18
* Clinical diagnosis of subaortic stenosis and underwent surgery

Exclusion Criteria:

* Diagnosed with hypertrophic cardiomyopathy
* Underwent concomitant previous surgical repair for aortic valve or SAS
* Follow-up time less than 1 year or lack of detailed information.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients age from 0-18 underwent SAS surgical repair at Fuwai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of Postoperative significant AR (SAR) | Through study completion, an average of 4 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China